CLINICAL TRIAL: NCT03284268
Title: Phase I Study, Single Site, Open Label With Dose Escalation, for Evaluate Safety and the Oncolitic Adenovirus VCN-01 Activity in Patients With Refractory Retinoblastoma
Brief Title: Evaluate Safety and the Oncolitic Adenovirus VCN-01 Activity in Patients With Refractory Retinoblastoma
Acronym: RTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSJD-RTB-2015
Record Dates: First submitted 2017-08-17; First posted 2017-09-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Retinoblastoma, Recurrent
Keywords: Gene therapy
MeSH Terms: conditions — Retinoblastoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation of VCN-01 (Experimental): Dose lower : 2E+9 viral particules/eye Dose medium: 2E+10 viral particules/eye Dose high: 2E+11 viral particules/eye
  Interventions: Genetic: VCN-01

INTERVENTIONS:
Genetic: VCN-01 — VCN-01 intravitreal injection

SUMMARY:
Phase I study, single site, open label with dose escalation, for evaluate safety and the oncolitic Adenovirus VCN-01 activity in patients with refractory retinoblastoma.

DETAILED DESCRIPTION:
Phase I clinical trial, single-center, open-label, dose-escalation study, to evaluate the safety of the VCN-01 and, secondarily, its anti-tumoral activity. The trial sample consists of approximately 13 patients aged between 1 and 12 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with retinoblastoma with a somatic mutation of the geneRB1 and active tumor in a single eye, or germinal mutation of RB1 with active tumor/s in an eye and the contralateral eye unaffected, enucleated or without tumor activity. In both cases, relapsed or refractory with the use of systemic, intraarterial or intravitreal chemotherapy or radiotherapy, in accordance with the availability at his/her referral site, in whom enucleation is the only recommended treatment under opinion of the medical team treating the case at the originating referral site.
2. Normal renal function: serum creatinine: <45μmol/L (0-2 years); <57μmol/L (3-6 years); <60μmol/L (7-10 years); <80μmol/L (11-13 years).
3. Normal Hepatic function: serum ALT: <0,52μkat/L (de 9 months -12 years); serum AST: 61-80 g/L (8 months - 5 years); 63-83 g/L (5-9 years); 63-82 g/L (9-12 years).
4. Adequate marrow reserve manifested in an absolute neutrophil count> 1000 / mm3, platelets> 100,000 / mm3 and hemoglobin> 8 g / dl, without transfusional or cytokine support at least one month prior to study entry.
5. Age greater than one year and less than 12 years at the time of inclusion in the study.
6. Informed consent form signed.

Exclusion Criteria:

1. Presence of factors that require immediate enucleation of the affected eye such as glaucoma, rubeosis iridis, anterior chamber involvement.
2. Comorbidities: Uncontrolled epilepsy with anticonvulsant treatment, cardiac disease not compensated by treatment.
3. Active Infections.
4. Other chronic or active acute diseases that under the criterion of the researcher were an exclusion criterion.
5. History of having received attenuated or live vaccines in the 30 days prior to inclusion in the study.
6. Any cause of Immunosuppression.
7. Trilateral Retinoblastoma.
8. Extraocular spread.
9. History of having received treatment for retinoblastoma with chemotherapy or radiation therapy by any means within 30 days prior to inclusion in the study.
10. Patients who can not complete the study procedures for reasons psychological or social.
11. Pregnancy. Female patients with procreative potential should be agree to undergo a blood or urine pregnancy test and the result should be negative to enter the study.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 180 days
  The safety and tolerability of two intravitreal injections of VCN-01 will be determined with dose escalation until the maximum tolerated dose (MTD) is established based on the evaluation of adverse events and the observation of any dose-limiting toxicity (TLD).

SECONDARY OUTCOMES:
Tumor response | 28 days
  Tumor response rate (ORR) to VCN-01 at 28 days post-administration.
VCN-01 | 180 days
  Virus presence in blood samples, aqueous humor, ocular surface and nasal swabs, and its difference between the viral particles before and after the treatment to evaluate the excretion profile of the CNV-01.
Immune response | 180 days
  The presence of neutralizing antibodies in blood samples in study patients to assess the immune response.

OTHER OUTCOMES:
Histopathology of enucleated eyes after treatment with VCN-01 | 180 days
  Presence of VCN-01 in vitreous humor samples of enucleated eyes

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Catalá Mora, Dr, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Anonymized individual data of participants will be shared with Authorities at the end of the Clinical development plan by the CTD (Common Technical Document). Results will be published in a scientific publication